CLINICAL TRIAL: NCT06218043
Title: An Iodine Balance Study in the Elderly
Brief Title: An Iodine Balance Study to Investigate the Recommended Iodine Intake in an Elderly Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenxing Guo (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Gansu Provincial Centre for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor-Investigator, Wenxing Guo, School of Public Health, Tianjin Medical University
Organization: Tianjin Medical University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 82204041-NSFC
Record Dates: First submitted 2023-12-27; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Nutrition, Healthy
Keywords: recommended intake of iodine; iodine balance study; thyroid diseases; elderly
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Intervention Model Description: When the first phase of the iodine balance study without intervention is completed. After an interval of 4 days, subjects who eat iodized salt will be included, the iodized salt will be replaced with non-iodized salt, and the second phase of the iodine balance experiment will begin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iodine intake intervention balance experiment (Other): Replace subjects' iodized salt with non-iodized salt.
  Interventions: Behavioral: Restrict subjects' intake of iodine-containing foods

INTERVENTIONS:
Behavioral: Restrict subjects' intake of iodine-containing foods — Replace subjects' iodized salt with non-iodized salt.

SUMMARY:
Current Chinese dietary iodine reference intake (DRIs) standards lack direct data on recommended iodine intake (RNI) in the elderly. The elderly have a high prevalence of thyroid diseases. The risk threshold of iodine intake in the elderly is unknown. Identifying the appropriate iodine intake for the elderly to maintain optimal thyroid function to reduce the burden on medical resources is a public health issue requiring high attention. The iodine balance study is an important method for exploring physiological iodine requirements. Few iodine balance studies have been conducted in the elderly. This study aimed to conduct an iodine balance study and provide information on the appropriate iodine intake level for elderly people.

DETAILED DESCRIPTION:
The investigators measured subjects' food and water intake throughout the day using weighing methods, and collected all urine and fecal samples. Food, drinking water, fecal and urine samples were taken to determine iodine concentrations. Each subject was required to participate in two phases of iodine balance studies. Each stage lasts 4 to 10 days. There was no intervention in the first half of the experiment, and there was an intervention of iodized salt/non-iodized salt consumption in the second half of the experiment. The appropriate level of iodine intake for the elderly was explored by fitting and analyzing the dose change relationship between iodine intake and iodine excretion.

ELIGIBILITY:
The target population of this study is elderly people over 60 years old. Adults living in the same household can also participate.

Inclusion Criteria:

1. aged 18 and above;
2. at least 5 years of local residence.

Exclusion Criteria:

1. family genetic diseases；
2. special dietary habits；
3. taking iodine-containing drugs or supplements；
4. metabolic diseases;
5. thyroid diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Iodine intake | Each phase of the iodine balance study lasts 4 to 10 days.
  Daily iodine intake includes dietary iodine intake and drinking water iodine intake.
Iodine excretion | Each phase of the iodine balance study lasts 4 to 10 days.
  Daily iodine excretion includes urinary iodine excretion and fecal iodine excretion.

SECONDARY OUTCOMES:
thyroid function indexes | Within one week before the start of the experiment.
  FT3、FT4、TSH、TPOAb、TGAb. Each subject was asked to collect venous blood twice (before the experiment and within one week after the intervention) to measure indicators of thyroid work.
thyroid volumn | Within one week before the start of the experiment.
  Thyroid volume was measured using thyroid B-ultrasound.
salivary iodine | 4 to 10 days
  Every time the subject urinates, 2ml of saliva is collected.
blood pressure | Within one week before the start of the experiment.
  Subjects had their blood pressure measured before and after the study.
fasting blood glucose | Within one week before the start of the experiment.
  Subjects had their fasting blood glucose measured before and after the study.

CONTACTS AND LOCATIONS:
Overall Officials: Wenxing Guo, Study Chair — Department of Nutrition and Food Hygiene, School of Public Health, Tianjin Medical University
Locations (3):
- China (3):
  - Gansu provincial center for disease control and prevention, Lanzhou, Gansu
  - Shandong provincial institute for endemic disease control, Jinan, Shandong
  - Tianjin Medical University, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
The data of the study are available from the project leader upon reasonable request.

REFERENCES:
- [Background] Zimmermann MB, Boelaert K. Iodine deficiency and thyroid disorders. Lancet Diabetes Endocrinol. 2015 Apr;3(4):286-95. doi: 10.1016/S2213-8587(14)70225-6. Epub 2015 Jan 13. PMID 25591468
- [Background] Farebrother J, Zimmermann MB, Andersson M. Excess iodine intake: sources, assessment, and effects on thyroid function. Ann N Y Acad Sci. 2019 Jun;1446(1):44-65. doi: 10.1111/nyas.14041. Epub 2019 Mar 20. PMID 30891786
- [Background] Dold S, Zimmermann MB, Baumgartner J, Davaz T, Galetti V, Braegger C, Andersson M. A dose-response crossover iodine balance study to determine iodine requirements in early infancy. Am J Clin Nutr. 2016 Sep;104(3):620-8. doi: 10.3945/ajcn.116.134049. Epub 2016 Jul 27. PMID 27465383
- [Background] Malvaux P, Beckers C, De Visscher M. Iodine balance studies in nongoitrous children and in adolescents on low iodine intake. J Clin Endocrinol Metab. 1969 Jan;29(1):79-84. doi: 10.1210/jcem-29-1-79. No abstract available. PMID 5762324
- [Background] Ingenbleek Y, Malvaux P. Iodine balance studies in protein-calorie malnutrition. Arch Dis Child. 1974 Apr;49(4):305-9. doi: 10.1136/adc.49.4.305. PMID 4208456
- [Background] Chinese Nutrition Society. Chinese Dietary Reference Intakes. Beijing, People's Medical Publishing House. 2014: 230-237. Chinese.
- [Background] Yang L, Wang J, Yang J, Zhang H, Liu X, Mao D, Lu J, Gu Y, Li X, Wang H, Xu J, Tan H, Zhang H, Yu W, Tao X, Fan Y, Cai Q, Liu X, Yang X. An iodine balance study to explore the recommended nutrient intake of iodine in Chinese young adults. Br J Nutr. 2020 Dec 14;124(11):1156-1165. doi: 10.1017/S0007114520002196. Epub 2020 Jun 22. PMID 32624007
- [Background] Tan L, Tian X, Wang W, Guo X, Sang Z, Li X, Zhang P, Sun Y, Tang C, Xu Z, Shen J, Zhang W. Exploration of the appropriate recommended nutrient intake of iodine in healthy Chinese women: an iodine balance experiment. Br J Nutr. 2019 Mar 14;121(5):519-528. doi: 10.1017/S0007114518003653. Epub 2018 Dec 11. PMID 30526700